CLINICAL TRIAL: NCT04058626
Title: Comparative Diagnostic Accuracy Study of Bedside Tests Used to Detect Arterial Disease in Diabetes:
Brief Title: TEsting for Arterial Disease in Diabetes (TrEAD) Study
Status: Completed | Type: Observational
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 17HH4091
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Results first posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Diabetic Foot; Peripheral Arterial Disease; Diabetic Foot Ulcer; Peripheral Vascular Diseases; Peripheral Artery Disease; Critical Limb Ischemia; Critical Lower Limb Ischemia
Keywords: Peripheral Vascular Diseases; Diabetic Foot; Critical Limb Ischemia; Diagnosis; Peripheral arterial disease; Diabetic foot ulcer; Duplex ultrasound; Ultrasound
MeSH Terms: conditions — Diabetic Foot; Peripheral Arterial Disease; Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia; Disease | interventions — Ankle Brachial Index

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transcutaneous pressure of oxygen (TcPO2) — Measurements will be taken from the dorsum of the foot using an automated machine equipped with Clark electrodes.
Diagnostic Test: Toe Brachial Pressure Index (TBPI) — TBPI will be measured using the photoplethysmography (PPG) method, employing an infrared sensor placed on the hallux and index finger.
Diagnostic Test: Podiatry Ankle Duplex scan (PAD-scan) — Podiatry ankle duplex scan (PAD-scan) involves using an ultrasound machine to visualise the anterior and posterior tibial arteries at the ankle.
Diagnostic Test: Duplex Assist — Continuous Doppler device which gives visual display of arterial spectral waveform at the ankle.
Diagnostic Test: Ankle Brachial Pressure Index (ABPI) — A sphygmomanometer-cuff placed at the ankle and a handheld continuous wave Doppler device will be used to measure the systolic pressure of the DPA and PTA.

SUMMARY:
This study will focus on determining;

* How accurate the test is in detecting poor circulation
* How it's accuracy compares to other commonly used tests, and
* Whether test results are linked to the chance of ulcer healing or amputation. Across 2 hospitals, 305 diabetic patients will be scanned using the focused ultrasound test as well as other commonly used tests to detect poor circulation. Their results will be compared to a full version of the ultrasound test to identify the most accurate.

DETAILED DESCRIPTION:
In the UK, over 7,000 amputations are performed each year because of diabetes. Most of these (80%) occur when a foot wound, also known as an ulcer, does not heal. The most important cause of this is poor circulation to the feet. Currently, there are no accurate tests that foot specialists can use to detect poor circulation when they see patients. Because of this, poor circulation can be missed and its treatment delayed.

A focused ultrasound test at the ankle, using a sensor and gel on the skin, can detect poor circulation. It is safe, painless and I have previously proven that it can be learned and performed quickly. It may help avoid amputations by detecting poor circulation so that it can be treated quickly.

ELIGIBILITY:
Inclusion Criteria:

* All diabetic patients presenting to the diabetic foot clinics will be eligible for the study.

Exclusion Criteria:

* Patients unable to provide informed consent will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred to the diabetic foot clinics at these sites will be asked to take part in the study.
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-10-18 (Actual); Study Completion 2019-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer Usman, Principal Investigator — Imperial College London
Locations (2):
- United Kingdom (2):
  - West Middlesex University Hospital, London
  - Imperial College NHS Healthcare Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elghazaly H, Howard T, Sanjay S, Mohamed OG, Sounderajah V, Mehar Z, Davies AH, Jaffer U, Normahani P. Evaluating the prognostic performance of bedside tests used for peripheral arterial disease diagnosis in the prediction of diabetic foot ulcer healing. BMJ Open Diabetes Res Care. 2023 Mar;11(2):e003110. doi: 10.1136/bmjdrc-2022-003110. PMID 36918215
- [Derived] Normahani P, Poushpas S, Alaa M, Bravis V, Aslam M, Jaffer U. Study protocol for a comparative diagnostic accuracy study of bedside tests used to detect arterial disease in diabetes: TEsting for Arterial disease in Diabetes (TrEAD) study. BMJ Open. 2020 Feb 5;10(2):e033753. doi: 10.1136/bmjopen-2019-033753. PMID 32029491

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Participants: Participants with diabetes were consecutively enrolled into the study across 2 centers.
Period: Overall Study
Arm/Group | Study Participants
Started | 305
Completed | 305
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Participants
Number analyzed (Participants) | 305
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 72 [62 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99
  Male | 206
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Active ulceration [Count of Participants; unit: Participants] | 123
Neuropathy [Count of Participants; unit: Participants] | 203

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy
Description: Diagnostic accuracy of the PAD-scan and other bedside tests will be compared to the results of a full lower limb Duplex Ultrasound scan (reference test).
Time Frame: 1 hour; all tests will be performed on the same day of presentation.
Population: Missing data were observed in 7 (2.3%) patients for ABPI, 71 (23.3%) patients for TBPI and 16 (5.2%) patients for TcPO2.
Measure: Number (95% Confidence Interval); unit: Percent
Arm/Group | Study Participants
Number analyzed (Participants) | 305
Percent
  PAD-scan sensitivity | 95 [90 to 97]
  PAD-scan specificity | 77 [67 to 84]
  TBPI sensitivity: number analyzed (Participants) | 234
  TBPI sensitivity | 60 [51 to 68]
  TBPI specificity: number analyzed (Participants) | 234
  TBPI specificity | 86 [77 to 92]
  Pulse sensitivity | 43 [36 to 50]
  Pulse specificity | 81 [72 to 88]
  Doppler (audible) sensitivity | 74 [67 to 80]
  Doppler (audible) specificity | 76 [66 to 84]
  Doppler (visual) sensitivity | 83 [77 to 88]
  Doppler (visual) specificity | 75 [65 to 83]
  ABPI sensitivity: number analyzed (Participants) | 298
  ABPI sensitivity | 60 [53 to 67]
  ABPI specificity: number analyzed (Participants) | 298
  ABPI specificity | 75 [66 to 83]
  TcPO2 sensitivity: number analyzed (Participants) | 289
  TcPO2 sensitivity | 31 [24 to 38]
  TcPO2 specificity: number analyzed (Participants) | 289
  TcPO2 specificity | 79 [69 to 86]

ADVERSE EVENTS:
Time Frame: The study duration is short and transient as index and reference tests are completed in a single visit. Study duration is therefore less than 1 hour. Additionally, all tests were non-invasive. Therefore, adverse events were not foreseen or encountered.
Arm/Group | Study Participants
All-Cause Mortality (participants affected / at risk) | 0/305
Serious Adverse Events (participants affected / at risk) | 0/305
Other Adverse Events (participants affected / at risk) | 0/305

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT04058626/Prot_SAP_000.pdf